CLINICAL TRIAL: NCT02478307
Title: Mechanisms of Mindfulness Meditation, Cognitive Therapy, and Mindfulness-Based Cognitive Therapy for Low Back Pain
Brief Title: Coping Skills Training for Living With Chronic Low Back Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: University of Washington (Other); University of Alabama at Birmingham (Other); Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Dr Melissa Day, NHMRC Early Career Fellow, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UQueensland
Record Dates: First submitted 2015-06-09; First posted 2015-06-23 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Low Back Pain
Keywords: chronic low back pain; mindfulness meditation; cognitive therapy; mindfulness-based cognitive therapy; efficacy; mechanisms; coping
MeSH Terms: conditions — Low Back Pain | interventions — Cognitive Behavioral Therapy; Mindfulness; Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive Therapy (Active Comparator): Eight, 2-hours sessions of group delivered cognitive therapy.
  Interventions: Other: Cognitive Therapy
- Mindfulness Meditation (Active Comparator): Eight, 2-hours sessions of group delivered mindfulness meditation.
  Interventions: Other: Mindfulness Meditation
- Mindfulness-Based Cognitive Therapy (Active Comparator): Eight, 2-hours sessions of group delivered mindfulness-based cognitive therapy
  Interventions: Other: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Other: Cognitive Therapy
  Arms: Cognitive Therapy
Other: Mindfulness Meditation
  Arms: Mindfulness Meditation
Other: Mindfulness-Based Cognitive Therapy
  Arms: Mindfulness-Based Cognitive Therapy

SUMMARY:
Up to 80% of Australians experience back pain and 10% have significant disability as a result. There is a critical need for the development and evaluation of innovative treatments that have the capacity to target the multidimensional nature of chronic low back pain. This study will compare the effects and mechanisms of Mindfulness Meditation, Cognitive Therapy, and Mindfulness-Based Cognitive Therapy for chronic low back pain. Results will ultimately lead to streamlined interventions designed to efficiently maximise benefit.

DETAILED DESCRIPTION:
Up to 80% of Australians experience back pain and 10% have significant disability as a result. This translates into substantial economic cost with far reaching psychological, emotional and social implications. Unfortunately, the treatment options for chronic low back pain (CLBP) are limited and typical medical/pharmacological approaches entail potentially serious side-effects (e.g., opioid addiction). There is a critical need for the development and evaluation of innovative interventions that have the capacity to target the multidimensional nature of CLBP.

Research indicates that psychosocial interventions for CLBP are viable treatment approaches that entail few (if any) deleterious side effects and can have benefit beyond pain reduction. Cognitive Therapy (CT) and Mindfulness Meditation (MM) have both been found to be feasible and effective for CLBP. A promising recently developed treatment that combines aspects of CT and MM is Mindfulness-Based Cognitive Therapy (MBCT). MBCT has been successfully applied to problems such as depression and headache; however, this approach has not been investigated for CLBP.

Thus, the current study is a randomised controlled trial (RCT) designed to examine the effects and mechanisms (i.e., how and for whom do these treatments work) of CT, MM, and MBCT for CLBP. Brain state data (electroencephalogram (EEG)) as well as self-report data will be examined to investigate the potential unique and shared mechanisms underlying treatment effects. Furthering the field's understanding of these treatments and their mechanisms will lead to the development of streamlined interventions designed to efficiently maximise benefit for individuals with CLBP, and that optimise relief from suffering.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Chronic pain of the low back (≥3 months) that is the primary source of reported pain
* Average pain intensity of ≥4 on a 10-point scale
* If currently taking analgesic or psychotropic medications, they must have been stabilised for ≥4 weeks prior to this study
* Be able to read, speak and understand English
* Be able to attend a weekly 2-hour therapy session for 8 concurrent weeks

Exclusion Criteria:

* Cognitive impairment, uncontrolled psychotic symptoms or current elevated suicidal ideation as this may interfere with group-delivered therapy (as evidenced by the 6-item screener)
* Chronic pain due to malignancy
* History of a medical condition that could produce an abnormal EEG and interfere with the tests of the effects of treatment on EEG (e.g., epilepsy, history of traumatic brain injury)
* Currently receiving other psychosocial pain treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Pain interference PROMIS scale | pre to post-treatment (at least 8 weeks)
  Participants are assessed pre-treatment and then following the 8-week treatment (post-treatment); change in pain interference is assessed via the PROMIS scale

SECONDARY OUTCOMES:
Pain intensity assessed via the numerical rating scale (NRS) | pre to post-treatment (at least 8 weeks)
  Participants are assessed pre-treatment and then following the 8-week treatment (post-treatment); change in pain intensity is assessed via the numerical rating scale (NRS)
Pain catastrophizing assessed via the Pain Catastrophizing Scale | pre to post-treatment (at least 8 weeks)
  Participants are assessed pre-treatment and then following the 8-week treatment (post-treatment); change in pain catastrophizing is assessed via the Pain Catastrophizing Scale
Mindfulness assessed via the FFMQ | pre to post-treatment (at least 8 weeks)
  Participants are assessed pre-treatment and then following the 8-week treatment (post-treatment); change in mindfulness is assessed via the FFMQ
Pain acceptance assessed via the CPAQ | pre to post-treatment (at least 8 weeks)
  Participants are assessed pre-treatment and then following the 8-week treatment (post-treatment); change in pain acceptance is assessed via the CPAQ
Psychological functioning PROMIS scale | pre to post-treatment (at least 8 weeks)
  Participants are assessed pre-treatment and then following the 8-week treatment (post-treatment); change in psychological functioning is assessed via the PROMIS scale
Emotional functioning PROMIS scale | pre to post-treatment (at least 8 weeks)
  Participants are assessed pre-treatment and then following the 8-week treatment (post-treatment); change in emotional functioning is assessed via the PROMIS scale
Physical functioning PROMIS scale | pre to post-treatment (at least 8 weeks)
  Participants are assessed pre-treatment and then following the 8-week treatment (post-treatment); change in physical functioning is assessed via the PROMIS scale
Delta, theta, alpha, beta, and gamma bands assessed via EEG | pre to post-treatment (at least 8 weeks)
  Participants are assessed pre-treatment and then following the 8-week treatment (post-treatment); change in brain state data is assessed via EEG

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Day, MA(Clin), PhD, Principal Investigator — The University of Queensland
Locations (1):
- The University of Queensland, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Day MA, Matthews N, Newman A, Mattingley JB, Jensen MP. An evaluation of the behavioral inhibition and behavioral activation system (BIS-BAS) model of pain. Rehabil Psychol. 2019 Aug;64(3):279-287. doi: 10.1037/rep0000274. Epub 2019 Mar 28. PMID 30920244